CLINICAL TRIAL: NCT02291835
Title: Dietary Intakes and Periodontal Outcomes After Sanative Therapy
Status: Completed | Type: Observational
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor and Canada Research Chair in Bone and Muscle Development, Brock University
Other Study IDs: BrockU
Record Dates: First submitted 2014-10-16; First posted 2014-11-17 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Periodontitis is a chronic inflammatory disease and a significant risk factor for tooth loss. While a link between diet and periodontal health exists, the relationship between diet and healing following periodontal therapy has yet to be investigated.The objective of this study was to determine if higher intakes of foods and nutrients with antioxidant or anti-inflammatory activity are associated with reduced probing depth following sanative therapy. Sanative therapy is a first line cost-effective treatment to manage periodontal disease and thus prevent tooth loss. Patients with chronic generalized periodontitis undergoing sanative therapy were recruited for the study. Mean probing depth was assessed at baseline and 8-16 weeks following sanative therapy. Dietary intakes of fruits, vegetables, vitamins and dietary fats were estimated using the Block 2005 food frequency questionnaire and supplement use was recorded using a questionnaire. A small venous blood sample was also collected at baseline to measure serum 25-hydroxyvitamin D concentrations.

DETAILED DESCRIPTION:
Oral health, specifically the retention of teeth, is inextricably and positively linked with nutritional status of an individual. The emerging inter-relationships among obesity, type II diabetes metabolic syndrome, acute coronary syndrome and/or breast cancer with the etiology of periodontal disease identify nutrition as having a unique role in potentially modulating these complex relationships. Some nutrients such as vitamin D and fatty acids have been studied more extensively than other nutrients. Cross-sectional studies using National Health and Nutrition Examination Survey (NHANES) data or other cohorts have identified that individuals with higher intakes of vitamin D or omega-3 polyunsaturated fatty acids have a decreased risk of periodontal disease and tooth loss. One study has identified that individuals with better vitamin D status (measured as serum 25-hydroxyvitamin D) have better recovery after sanative therapy. Sanative therapy is a routine, first line cost-effective treatment to manage periodontal disease and thus prevent tooth loss. It is a non-surgical process involving mechanical debridement of bacterial biofilms on the roots of teeth, below the level of the gum line. Although one study has reported associations between vitamin D and outcomes after sanative therapy, the status of other nutrients or overall dietary patterns has not been assessed in relation to recovery from sanative therapy. The objective of this study was to determine if higher intakes of foods and nutrients with antioxidant or anti-inflammatory activity, including fruits, vegetables, β-carotene, vitamin C, vitamin D, vitamin E and omega-3 fatty acids were associated with reduced probing depth following sanative therapy.

The study took place at a periodontal clinic in Southern Ontario, Canada. Prior to enrolment, patients attended a consultation where a baseline periodontal examination, including measurement of probing depth at six sites per tooth was completed. Patients with chronic generalized periodontitis who were then prescribed sanative therapy as part of their treatment plan were invited to participate in the study. The study was explained to them and they were presented with a letter of invitation. Written consent was then obtained from patients wishing to participate.

Patients returned to the clinical approximately two months later for their sanative therapy appointment. Prior to meeting with the hygienist who performed sanative therapy, participants met with a study nurse. The nurse collected a venous blood sample, which was used for measurement of serum 25-hydroxyvitamin D concentrations. The nurse also measured participant's height, weight, waist circumference and hip circumference. After sanative therapy was performed, participants were provided with the Block Food Frequency Questionnaire and a supplement use questionnaire to be completed at home. Participants then returned to the clinic 8 -16 weeks later for their routine follow-up examination, which included measurement of periodontal probing depth. Additionally, information including participants age, sex, health conditions, medications, allergies and smoking habits was recorded from the medical forms that were completed during their consultation visit.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing sanative therapy were eligible.

Exclusion Criteria:

* under 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing sanative therapy for the treatment of chronic generalized periodontitis.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Periodontal healing evaluated based on changes in mean probing depth | Baseline and between 8 and 16 weeks after sanative therapy
  Healing is evaluated based on changes in mean probing depth

OTHER OUTCOMES:
Dietary nutrient intakes | Completed by participant anytime between study enrolment and follow-up (8 to 16 weeks after sanative therapy)
  Dietary intakes were measured using the BLOCK food frequency questionnaire
Supplemental nutrient intakes | Completed by participant anytime between study enrolment and follow-up (8 to 16 weeks after sanative therapy)
  Supplemental intakes were measured using a dietary supplement use questionnaire
Serum 25-hydroxyvitamin D concentrations | Sample collected at baseline visit when sanative therapy was performed
  A venous blood sample was collected and sent to a medical laboratory for vitamin D testing.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy E Ward, PhD, Principal Investigator — Professor

REFERENCES:
- [Derived] Dodington DW, Fritz PC, Sullivan PJ, Ward WE. Higher Intakes of Fruits and Vegetables, beta-Carotene, Vitamin C, alpha-Tocopherol, EPA, and DHA Are Positively Associated with Periodontal Healing after Nonsurgical Periodontal Therapy in Nonsmokers but Not in Smokers. J Nutr. 2015 Nov;145(11):2512-9. doi: 10.3945/jn.115.211524. Epub 2015 Sep 30. PMID 26423734